CLINICAL TRIAL: NCT04561843
Title: 3D Transperineal Ultrasound of the Pelvic Floor Muscles in Women With Pelvic Floor Disorders: A Cross-sectional Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sief el eslam Ahmed Ali, Principal Investigator, Assiut University
Other Study IDs: AUG2020
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: Women complaining of any of the pelvic floor disorder symptoms such as: Pelvic organ prolapse (POP), Stress urinary incontinence (SUI), urgency symptoms of obstructed defecation, fecal incontinence (FI), pelvic pain, and/or sexual problems.
  Interventions: Diagnostic Test: pelvic floor ultrasound
- control group: Women not complaining of any of the pelvic floor disorder symptoms
  Interventions: Diagnostic Test: pelvic floor ultrasound

INTERVENTIONS:
Diagnostic Test: pelvic floor ultrasound — 2D and 3D trans-perineum ultrasound examinations will be performed by single examiner who was blind to clinical data, using a GE Voluson 730 machine (GE Medical System Kretz Technik, Zipf, Austria) with a RAB 4-8 MHz curved array volume transducer. In the supine position, with flexed and slightly abducted hips after urine voiding. The transducer was placed on the perineum, in the mid sagittal plane with minimal pressure being applied after covering it with an un-powdered glove or thin plastic wrap for hygienic reasons

SUMMARY:
The present study aimed to evaluate the levator ani muscle in both morphology (rest), and function (contraction and valsalva) in symptomatic women using 2D, 3D trans-perineum ultrasound (TPUS), to compare these features to clinical digital palpation and symptoms, and helping in diagnosis of muscle dysfunction.

DETAILED DESCRIPTION:
The prevalence of Pelvic floor dysfunction is high, affecting millions of women worldwide in different conditions (social, sexual, physical, psychological, domestic relationships, financial, etc.), many people still have no, limited knowledge, or awareness of pelvic floor health and so do not have, or seek how to prevent or correct these disorders . This dysfunction may be presented as pelvic organ prolapse, stress urinary incontinence, fecal incontinence , chronic pelvic pain, sexual problems, and/or chronic constipation . Assessment of pelvic floor muscle activity plays a major role in Urogynecology and physiotherapy as a part of the conservative treatment of pelvic floor disorders (PFD) . Presence of Levator avulsion is a major risk factor for female pelvic organ prolapse (POP) and recurrence after surgical correction . This dysfunction can be diagnosed clinically using vaginal palpation . Palpation is subjective, less reproducible, and difficult to teach than imaging methods [6]. Studies that used ultrasound for assessment of pelvic floor muscle activity and strength are still few . The present study aimed to evaluate the levator ani muscle in both morphology (rest), and function (contraction and valsalva) in symptomatic women using 2D, 3D trans-perineum ultrasound (TPUS), to compare these features to clinical digital palpation and symptoms, and helping in diagnosis of muscle dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Women complaining of any of the pelvic floor disorder symptoms.

Exclusion Criteria:

* women with a history of chronic intestinal disease (Crohn's disease, ulcerative colitis), acute gastroenteritis within the week preceding consultation women who underwent any surgical or diagnostic procedure involving the anal canal

Ages: 21 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female
Study Population: Women complaining of any of the pelvic floor disorder symptoms such as: Pelvic organ prolapse (POP), Stress urinary incontinence (SUI), urgency symptoms of obstructed defecation, fecal incontinence (FI), pelvic pain, and/or sexual problems.
Sampling Method: Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
pelvic floor muscle function. | 15 miutes
  The hiatal antro-posterior distance (LHap) between the inferior margin of the pubic symphysis and the pubo-rectalis sling was measured at rest, on maximum contraction, and at valsalva. The percentage difference decrease [valuerest valuecontraction/ valuerest] for contraction is calculated as a measurement of pelvic floor muscle function.

IPD SHARING:
Plan to Share IPD: Undecided